CLINICAL TRIAL: NCT06456307
Title: Integration of Stepped Care for Perinatal Mood and Anxiety Disorders Among Women Attending MCH Clinics
Acronym: IPMH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kenyatta National Hospital (Other Government)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P425/04/2023; STUDY00017933 (Other: University of Washington); R01MH133266 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Depression, Anxiety; Antenatal Depression; Postnatal Depression
Keywords: perinatal mood and anxiety disorders; telepsychiatry; Problem management plus; Integrated Perinatal Mental Health; Pregnancy; Postpartum; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders; Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: A 1:1 cluster-randomized trial will be conducted in 20 facilities in Western Kenya among pregnant women (3rd trimester) with perinatal mood and anxiety (PMAD) symptoms (Patient Health Questionnaire-2 [PHQ-2]≥3 or Generalized Anxiety Disorder-7 [GAD-7]≥3). Control facilities will provide enhanced standard of care (PMAD screening followed by standard of care). Intervention facilities will provide IPMH. Effectiveness outcomes will be compared between study arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm: Enhanced Standard of care (No Intervention): Control facilities will provide enhanced standard of care. The enhanced standard of care will include two enhancements:
  1. HIV Testing Services (HTS) providers and lay workers will conduct screening for perinatal mood and anxiety disorders (PMAD) using the PHQ-2 and GAD-2.
  2. The study team will provide a PMAD referral information sheet to all control facilities describing inpatient and outpatient psychiatry services at the nearby referral hospitals
- Intervention arm: Integrated Perinatal Mental Health Program (IPMH) (Experimental): Intervention facilities will receive the Integrated Perinatal Mental Health Program (IPMH). This includes:
  1. Systematic screening for PMAD symptoms using PHQ-2 and GAD-2. Positive screeners (PHQ-2≥3 and/or GAD-2≥3) will then be referred to nurses to administer additional screening by PHQ-9 and GAD-7
  2. Non-specialist delivery of PM+ for participants with likely depression (PHQ-9≥10) or anxiety (GAD-7≥10) delivered weekly
  3. In-facility tele-linkage to mental health specialist for participants with severe depressive symptoms (PHQ-9≥15), those who endorse suicidality, or non-responders to Problem Management+
  Interventions: Behavioral: Integrated Perinatal Mental health program (systematic screening for PMAD, PM+ and tele-psychiatry)

INTERVENTIONS:
Behavioral: Integrated Perinatal Mental health program (systematic screening for PMAD, PM+ and tele-psychiatry) — The intervention includes systematic screening for PMAD symptoms using PHQ-2 and GAD-2, non-specialist delivery of PM+ for participants with likely depression (PHQ-9≥10) or anxiety (GAD-7≥10) and in-facility tele-linkage to mental health specialist for participants with severe depressive symptoms (PHQ-9≥15), those who endorse suicidality, or non-responders to PM+
  Arms: Intervention arm: Integrated Perinatal Mental Health Program (IPMH)

SUMMARY:
Perinatal mood and anxiety disorders (PMAD), defined as depression and anxiety during pregnancy or up to 1 year postpartum, account for substantial morbidity and mortality among birthing people globally especially in low- and middle-income countries. Several evidence-based interventions are recommended for identification and management of PMAD by non-specialist providers in resource-limited settings. This cluster-randomized trial seeks to evaluate the effect of a stepped-care intervention for screening and treatment of PMAD among perinatal women, on clinical and implementation outcomes.

DETAILED DESCRIPTION:
Globally, perinatal mood and anxiety disorders (PMAD) impacts 10-20% of perinatal women, with a pooled prevalence of depression at 11.9% and anxiety at 15.2%. Most of these cases go undetected and untreated since worldwide under 30% of those requiring mental health services have access to them. The Kenya Mental Health Action Plan 2021-2025 highlights a goal of expanding access to mental health services including in Maternal and Child Health clinics. In Kenya, over 95% of all pregnant women receive at least one antenatal care service from a skilled provider. However, mental health screening is not currently standardized in antenatal and postnatal care visits in Kenya, representing a missed opportunity to offer mental health services to those with PMAD symptoms.

Several evidence-based interventions are recommended by the WHO for identification and management of PMAD by non-specialist providers in resource-limited settings. However, their implementation in routine care in Kenya is currently limited, due to lack of provider training and comfort with perinatal mental health treatments and poor linkage across cadres of providers (such as primary care providers and mental health providers). Sustainable integration of perinatal mental healthcare in Kenya's routine perinatal services requires development and testing of tailored interventions that strengthen workforce capacity and facilitate linkage across provider cadres, as well as implementation strategies to facilitate high-quality intervention delivery. The investigators have identified three EBIs to promote perinatal mental health: universal WHO Mental Health Gap Action Programme (mhGAP)-recommended mental health screening, the Problem Management Plus (PM+) counseling intervention for women experiencing PMAD, and telepsychiatry for women with severe symptoms, suicidality or no response to PM+. The investigators propose to combine these interventions in a stepped care model, named the Integrated Perinatal Mental Health program (IPMH), and develop implementation strategies to support the model's integration into routine perinatal care in Kenya. The investigators will then evaluate IPMH's effectiveness and implementation outcomes in a Hybrid Type II trial. The study will be conducted in clinics in Kisumu, Siaya, and Homa Bay counties of Western Kenya, Kenya.

Broad objective: This study seeks to evaluate the effectiveness and implementation outcomes of Integrated Perinatal Mental Health Program (IPMH) that consists of universal mental health screening, problem management plus counseling intervention and telepsychiatry in a Hybrid Type II trial.

Aim 1: Using participatory design, optimize and adapt IPMH and develop implementation strategies.

Aim 2: Determine the effect of IPMH and implementation strategies on mental health, HIV care, and pregnancy outcomes among perinatal women from pregnancy to 6 months postpartum.

Aim 3: Determine effect of IPMH and its implementation strategies on service delivery and implementation outcomes, and identify multilevel drivers of successful implementation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant and ≥28 weeks gestation
* Attending ANC care at the facility
* ≥14 years old
* Screen positive for PMAD symptoms (PHQ-2≥3 and/or GAD-2≥3)
* Willing to return to the MCH and PMTCT clinic for study visits

Exclusion Criteria:

* Less than 28 weeks gestation
* Any woman at high risk of self-harm based on a study self-harm assessment protocol,
* Has cognitive impairments or psychotic symptoms

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2970 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Depression | 6-months postpartum
  Patient Health Questionnaire-9 (PHQ-9). Score range 0-27. Higher score indicates more severe depression symptoms; score ≥10 indicates symptoms of moderate-to-severe depression
Anxiety | 6-months postpartum
  Generalised Anxiety Disorder-7 item (GAD-7). Score range 0-21. Higher score indicates more severe anxiety symptoms; score ≥10 indicates symptoms of moderate-to-severe anxiety

SECONDARY OUTCOMES:
Quality of life | 6-months postpartum
  World Health Organisation Quality-of-Life Brief Version (WHOQOL-BREF) score. Score range 0 - 100. Higher scores indicate higher quality of life.
Adverse pregnancy outcomes | 6-weeks postpartum
  Any adverse pregnancy outcomes defined as the following: Pregnancy loss, stillbirth, pre-term birth, low birth weight, intrauterine growth restriction, neonatal hospital admission and neonatal death
Mechanism of action for PM+ (use of behavioral and psychosocial coping skills) | 6-weeks postpartum
  Reducing Tension Checklist. Score range 0 - 40. Higher score indicates more use of behavioral and psychosocial coping skills.

CONTACTS AND LOCATIONS:
Overall Officials: John Kinuthia, MBChB, MMed, MPH, Principal Investigator — Kenyatta National Hospital; Keshet Ronen, MPH, PhD, Principal Investigator — University of Washington; Amritha Bhat, MBBS, MD, MPH, Principal Investigator — University of Washington
Locations (2):
- Kenya (2):
  - Kenyatta National Hospital, Nairobi
  - HomaBay, Siaya and Kisumu, Western Kenya

IPD SHARING:
Plan to Share IPD: Yes
Data from IPMH will be available through the NMIH Data Archive
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: At the end of the project.
Access Criteria: The NIH will provide access to scientific investigators for research purposes. Qualified researchers who have completed a Data Use Certification and received approval from the NDA Data Access Committee (DAC) may be approved to access broadly shared data. A separate request process exists for access to data in federated sources. Additionally, the DAC and support staff at NIH have access to NDA shared data.